CLINICAL TRIAL: NCT07156045
Title: Clinical Study on the Safety and Efficacy of Anti-PSMA CAR NK Cells in Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC)
Brief Title: Study of Allogeneic Anti-PSMA CAR-NK Cell for Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, XINGNIANZENG, Vice President of the Hospital, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25/062-0062
Record Dates: First submitted 2025-08-07; First posted 2025-09-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer Castration-resistant Prostate Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Biological: anti-PSMA CAR-NK

INTERVENTIONS:
Biological: anti-PSMA CAR-NK — Targeting PSMA CAR-NK cells

SUMMARY:
At present, no cell drug with an indication for mCRPC has been approved for marketing in China, and there is no scholar to fight against it PSMA-CAR-NK cell therapy CRPC was reported in a study. Based on the previous basic research, our company has developed CAR-NK cell injection, hoping to further evaluate its safety, tolerability and preliminary efficacy in the treatment of mCRPC patients in clinical studies, and provide new possibilities for the selection of clinical treatment strategies

ELIGIBILITY:
Inclusion Criteria:

To enter the trial, subjects had to meet all of the following eligibility criteria:

1. diagnosed metastatic castration-resistant prostate cancer (mCRPC);
2. Castration level of serum testosterone (< 50 ng/dL or < 1.7 nmol/L);
3. Positive expression of PSMA;
4. According to the definition of CRPC in the Guidelines for the Diagnosis and Treatment of Prostate Cancer (2022 edition), the disease still progresses after castration and meets any of the following criteria:

   A.According to the increase in PSA level, there should be 3 consecutive increases in PSA at least 1 week apart (the increase in PSA is more than 50% of the minimum value, and PSA > 2 ng/mL); B.Progression of bone disease as defined by PCWG3, defined as the presence of 2 or more new lesions on bone scan; C.CT or MRI results suggested measurable metastasis (lymph node short diameter > 15 mm was defined as lymph node metastasis as assessed by RECIST 1.1);
5. Expected survival time ≥6 months;
6. Toxicity of any previous treatment had recovered to ≤ grade 1 at the time of enrollment (except hair loss and hearing loss);
7. ECOG score of patients 0-2;
8. Patients voluntarily participated and signed the informed consent, and followed the trial treatment plan and visit plan.

Exclusion Criteria:

Subjects who meet one of the following conditions will not be enrolled in the trial:

1. Previous recipients of other cell therapy products, such as dendritic cells (DC), multiple cytokine-induced killer cells (CIK), T cells, natural killer cells (NK), chimeric antigen receptor T-cell immunotherapy (CAR-T), etc.;
2. Patients with a history of biological macromolecule drug allergy;
3. Abnormal function of major organs:

   A. Neutrophil count (ANC) < 1.5×109/L; Platelet count (Plt) < 100×109/L; Hemoglobin (Hb) < 9 g/dL; B. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥2.5×ULN (≥5×ULN for liver metastases); C. Renal function: serum creatinine (Cr) ≥1.5×ULN; D. Prothrombin time (PT) > 15 s, activated partial thrombin time (APTT) was prolonged or shortened by more than 10 s (normal reference value 23 s-37 s), or international normalized ratio (INR) > 1.7; E. Pulmonary function: Severe respiratory diseases (active pulmonary tuberculosis, chronic obstructive pulmonary disease, interstitial lung disease, etc.)
4. Previous treatment with any PSMA-targeted therapy;
5. active autoimmune diseases (including connective tissue disease, uveitis, sarcoidosis, inflammatory bowel disease, or multiple sclerosis) or need long-term immunosuppressive therapy of severe autoimmune disease (screening clinic within six weeks before any immunosuppressive therapy), or by the researchers determine in 3 months will be recurrence of subjects;
6. have had other malignancies other than prostate cancer (other than basal or squamous cell skin cancer) in the past 5 years that are currently clinically significant and require intervention;
7. Any active (viral, bacterial, fungal) infection currently being treated or any infection requiring intravenous antibiotics for 7 or more days or intervals during the past 6 weeks or any active infection requiring oral antibiotics during the past 1 week;
8. untreated chronic active hepatitis B, or chronic hepatitis B virus carriers with HBV DNA≥1000 copies /mL, or active hepatitis C patients;
9. Patients who have participated in other clinical trials and used study drugs within 3 months;
10. Effective contraceptive measures cannot be adopted ;
11. In the opinion of the investigator, there are other factors that are not suitable for inclusion or affect the participant's participation or completion of the study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment related adverse events as assessed by CTCAE v5.0 | Baseline to 1 year post infusion
  Defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment

SECONDARY OUTCOMES:
The pharmacokinetic analysis of Anti-PSMA CAR-NK Cell | D0, D1, D3, D7, D8, D10, D14, D15, D17, D28±1, D60±2, D120±2, D180±7, D270±7, and D365±7 post infusion
  Changes in the number of CD56+/ CD3 Anti-PSMA CAR-NK Cell in peripheral blood over time
The pharmacodynamics analysis of Anti-PSMA CAR NK Cell | Baseline to infusion date, D28±1, D60±2, D120±2, D180±7, D270±7, and D365±7
  Changes of total prostate specific antigen (tPSA) and free prostate specific antigen (fPSA) in peripheral blood
The proportion of patients with a decrease in PSA levels from baseline | Baseline to D28±1, D60±2, D120±2, D180±7, D270±7, and D365±7 post infusion
  PSA response rate
Progression-free survival (PFS) after Anti-PSMA CAR NK Cell infusion | Baseline to 1 year post infusion
  Survival time of patients
Time to clinical progression | Baseline to D28±1, D60±2, D120±2, D180±7, D270±7, and D365±7 post infusion
  The time from baseline to the appearance of increased PSA levels or imaging progression.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China